CLINICAL TRIAL: NCT07185386
Title: Effects of a Dietary Supplement Composed of Diosmin, Hesperidin, Bromelain, and Ruscus Aculeatus on the Quality of Life in Subjects With Lower Limb Disorders Possibly Prodromal to Chronic Venous Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ekalab S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VSV-25-001
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Prodromal to Chronic Venous Disease
MeSH Terms: interventions — Hesperidin; Bromelains

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VESVEIN (Experimental): VESVEIN Gambe, (Ekalab S.r.l., Italia)
  Interventions: Dietary Supplement: combination of diosmin, hesperidin, bromelain, and Ruscus aculeatus (Vesvein Gambe)

INTERVENTIONS:
Dietary Supplement: combination of diosmin, hesperidin, bromelain, and Ruscus aculeatus (Vesvein Gambe) — Although there is extensive clinical and pharmacological evidence regarding the activity of the individual components of the product, the specific effect of the fixed combination of diosmin, hesperidin, bromelain, and Ruscus aculeatus as a single entity on quality of life in subjects with symptoms compatible with the early stages of Chronic Venous Disease (CVD) has not yet been explored.

SUMMARY:
The primary objective of the study is to evaluate, after 12 weeks (visit 3, V3), the effect of the combination of diosmin, hesperidin, bromelain, and Ruscus aculeatus (Vesvein Gambe) on any changes in the total quality of life score, measured using the CIVIQ-20 (Chronic Venous Insufficiency Quality of Life Questionnaire), compared to baseline (visit 1, V1), in individuals with subjective symptoms in one or both lower limbs attributable to Chronic Venous Disease (CVD).

ELIGIBILITY:
Inclusion Criteria:

* Both sexes;
* Age ≥18 years;
* Signed informed consent form for participation in the study;
* Presence of at least one clinical symptom possibly related to chronic venous disease (such as heaviness and/or swelling and/or pain in the lower limbs, nighttime cramps, tired/heavy legs, itching, burning and/or warmth, tingling, or restlessness in the lower limbs);
* Willingness to participate in the study and to comply with the study procedures, as confirmed by signing the written informed consent.

Exclusion Criteria:

Pregnancy or current breastfeeding; Women of childbearing potential who are not using adequate birth control methods (either hormonal contraception in the form of contraceptive pills, or barrier birth control methods used in combination with a spermicidal product such as foam, gel, or film).

[For the entire duration of the study, women of childbearing potential-defined as those who are less than one year post-menopause or who have not undergone hysterectomy or tubal ligation-must use an effective method of contraception, in accordance with Note 3 of the ICH M3 Guideline. A contraceptive method is considered highly effective if it results in a failure rate of less than 1% per year. Effective contraceptive methods include: hormonal contraceptives containing estrogens and progestins (oral, intravaginal, transdermal) that inhibit ovulation; hormonal contraceptives containing progestins only (oral, injectable, implantable); intrauterine devices (IUDs); hormone-releasing intrauterine systems (IUS); partner vasectomy; sexual abstinence]; Individuals with chronic venous insufficiency classified as CEAP stages C3-C6 (see Annex 1); Individuals with a positive pitting edema sign detected at Visit 1 after signing the informed consent; Patients with documented deep vein thrombosis within the last 6 months; Current or recent (within the last 4 weeks) use of venoactive and/or anti-edematous products; Individuals scheduled for surgical procedures within 3 months of enrollment; Subjects with a history of heart failure (NYHA Class III-IV), chronic kidney disease, and/or severe hepatic insufficiency; Ongoing oncological or immunosuppressive diseases; Celiac disease; Drug and/or alcohol abuse; Neurological or psychiatric disorders that may impair the validity of informed consent and/or compromise adherence to the study procedures; Known allergy, hypersensitivity, or intolerance to any component of the investigational dietary supplement; Any medical or non-medical condition that, in the opinion of the Investigator, could interfere with the study or make participation unsafe; Subjects currently enrolled in other clinical trials, or who have received another investigational product within 30 days prior to study start; Individuals who have not signed the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Primary objective | 12 weeks
  The primary objective of the study is to evaluate after 12 weeks (visit 3, V3) the effect of the combination diosmin, hesperidin, bromelain and Ruscus aculeatus (Vesvein Legs) on any variations in the total quality of life score, measured using the questionnaire CIVIQ-20 (Chronic Venous Insufficiency Quality of Life Questionnaire) compared to baseline (visit 1, V1), in individuals with symptoms subjective to one or to both lower limbs and referable to Chronic Venous Disease (MVC).

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - AOU Policlinico Sant'Orsola Malpighi, Bologna, BO
  - Università degli Studi Magna Graecia, Catanzaro, CZ
  - IRCCS San Raffaele Pisana, Roma, Roma
  - Ospedale Policlinico Agostino Gemelli, Roma, Roma
  - Azienda ULSS7 Pademontana Regione Veneto, Bassano del Grappa, VI
  - Vi.Gi. Centro Polispecialistico, Vibo Valentia, VV

IPD SHARING:
Plan to Share IPD: Undecided